CLINICAL TRIAL: NCT07401537
Title: Efficacy and Safety of Extended-Dose Interval Immunotherapy Versus Standard-Dose Interval Immunotherapy for Advanced Triple-Negative Breast Cancer: A Multicenter Randomized Controlled Clinical Trial
Brief Title: Efficacy and Safety of Extended-Dose Interval Immunotherapy Versus Standard-Dose Interval Immunotherapy for Advanced Triple-Negative Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jieqiong Liu, M.D., Ph.D., Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYSKY-2025-962-02
Record Dates: First submitted 2026-01-17; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Triple -Negative Breast Cancer; Breast Cancer
Keywords: Immune-checkpoint inhibitors; Dose Interval
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extended-Dose Interval (Experimental): During the maintenance therapy phase, the dose of PD-1 inhibitors is consistent with that of the standard therapy phase, administered every 6 weeks (q6w); the dose of chemotherapy or TROP2-ADC drugs is consistent with that of the standard therapy phase, administered every 3 weeks (q3w).
  Interventions: Drug: Extended-Dose Interval Immunotherapy
- Standard-Dose Interval (Active Comparator): During the maintenance therapy phase, the dosages of PD-1 inhibitors, chemotherapy, or TROP2-ADC drugs are maintained at the same levels as those in the standard treatment phase, administered every 3 weeks (q3w).
  Interventions: Drug: Standard-Dose Interval Immunotherapy

INTERVENTIONS:
Drug: Extended-Dose Interval Immunotherapy — During the maintenance therapy phase, the dose of PD-1 inhibitors is maintained at the same level as in the standard treatment phase, with the dosing interval extended to every 6 weeks (q6w).
  Arms: Extended-Dose Interval
Drug: Standard-Dose Interval Immunotherapy — During the maintenance therapy phase, the dosage and dosing interval of PD-1 inhibitors are consistent with those in the standard therapy phase, administered every 3 weeks (q3w).
  Arms: Standard-Dose Interval

SUMMARY:
Triple-negative breast cancer (TNBC), defined by the lack of ER, PR and HER2 expression, is refractory to endocrine therapy and anti-HER2 agents. Chemotherapy was once the mainstay for advanced TNBC, but its limited efficacy necessitates optimized therapeutic strategies. TNBC's high TIL infiltration and elevated PD-L1 expression confer sensitivity to immune checkpoint inhibitors (ICIs), with ICI-chemotherapy combinations initially establishing first-line standard status. Emerging clinical evidence shows that ICI-antibody-drug conjugate (ADC) combinations outperform ICI-chemotherapy regimens, yet immune-related adverse events (irAEs) remain a critical clinical challenge. Expert consensus recommends continuing ICI therapy in advanced TNBC patients achieving CR, PR or SD after ICI-based combination therapy until disease progression or intolerable toxicity. Mechanistically, once ICIs reach target receptor saturation, dose escalation or high-frequency administration fails to boost efficacy but raises toxicity risk. Thus the investigators hypothesize that an ICI maintenance strategy with fixed dose and extended intervals can preserve efficacy, reduce toxicity, improve patient compliance, enhance quality of life and alleviate economic burden for advanced TNBC patients with CR/PR/SD after ICI-chemotherapy or ICI-ADC treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary consent to participate in this study and signing of the informed consent form.
2. The age of the signatory of the informed consent form should be ≥18 years old and ≤70 years old.
3. Advanced (locally recurrent inoperable or metastatic) TNBC confirmed by histology or cytology, defined as ER-negative, PR-negative, and HER2-negative.
4. PD-L1 IHC detection in tumor tissue with a CPS score ≥1.
5. Have received first-line standard immunotherapy combined with chemotherapy or immunotherapy combined with ADC and completed 6 cycles, with the last dose administered no more than 28 days before randomization.
6. The therapeutic efficacy was confirmed as CR, PR or SD after 6-cycle standard treatment according to the RECIST v1.1 criteria.
7. Plan to continue receiving immunotherapy.
8. An Eastern Cooperative Oncology Group performance-status score of 0 or 1.
9. The expected survival period exceeds 12 weeks.
10. Adequate organ function:.
11. No mental or intellectual abnormalities.
12. Willing and able to comply with the trial protocol during the trial period.
13. Female subjects of childbearing potential must agree to use highly effective contraceptive measures starting at least 7 days before the first dose and continuing until 24 weeks after the last dose. The serum pregnancy test result must be negative within 7 days prior to the first dose.

Exclusion Criteria:

1. Untreated active brain metastases or meningeal metastases.
2. Concomitant other malignant tumors with progression within the recent 5 years or requiring active treatment (excluding adequately treated and controlled carcinoma in situ and non-melanoma skin cancer).
3. Concomitant severe non-malignant diseases that would affect the patient's compliance or put the patient at risk.
4. Concomitant active infection.
5. Receiving other anti-tumor therapies or participating in other interventional clinical trials.
6. Inflammatory breast cancer.
7. Dementia, intellectual disability, or any mental disorders that hinder the understanding of the informed consent form.
8. History of allergic reactions to any components of the study drugs or existing contraindications to their use.
9. Presence of any active autoimmune diseases or history of autoimmune diseases.
10. Presence of poorly controlled clinical cardiac symptoms or diseases, such as:1) Heart failure of NYHA class II or above;2) Unstable angina pectoris;3) Myocardial infarction occurring within 1 year;4) Clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention.
11. Presence of grade ≥3 toxicities related to prior treatments that restrict the continuation of maintenance therapy.
12. History of immunodeficiency, including HIV positivity, active HBV/HCV infection, other acquired or congenital immunodeficiency diseases, and history of organ or allogeneic stem cell transplantation.
13. Vaccination with live vaccines within 4 weeks prior to the administration of study drugs or planned vaccination during the study period.
14. Prior administration of irinotecan, topotecan, or any other topoisomerase I inhibitors (including investigational topoisomerase I inhibitors), or known history of allergies to the above-mentioned drugs.
15. Use of systemic glucocorticoids at a dose exceeding 10 mg/day of prednisone equivalent within 14 days prior to the administration of study drugs, or planned long-term use of the above dose during the study period (topical, inhaled, or short-term (≤7 days) pulse doses ≤10 mg/day of prednisone equivalent, or physiological dose replacement therapy are allowed for inclusion).
16. Need for use of any immunosuppressants within 14 days prior to the administration of study drugs or planned use during the study period.
17. Pregnant or lactating women, or women of childbearing potential who refuse to accept contraceptive measures.
18. Patients who are difficult or impossible to follow up.
19. Subjects judged by the investigator to have conditions that may affect compliance or other circumstances making them unsuitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2025-12-31 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
mPFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years.
  Refers to the time from randomization date to the first observation of disease progression (based on RECIST v1.1 criteria) or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
mOS | From date of randomization until the date of death from any cause, assessed up to 3 years.
  The time from randomization date to any cause of death date.
DoR | From date of achieving CR or PR until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years.
  Refers to the time from the date of achieving CR or PR to the first disease progression (PD) or death from any cause, whichever occurs first.
DDC | From date of achieving CR, PR, or SD until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years.
  Refers to the time from the date of achieving CR, PR, or SD to the first evaluation as PD or death from any cause, whichever occurs first.
Assessment of quality of life via the EORTC QLQ-C30 questionnaire. | 3 years.
  Patient reported outcomes via the European Organisation for Research and Treatment of Cancer Core Quality of Life questionnaire (EORTC QLQ-C30). It contains 30 items and measures 5 functional scales (physical, role, emotional, cognitive, and social), a global health and quality of life scale, 3 symptom scales (fatigue, nausea/vomiting, and pain), and 6 single items (dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, and financial impact). The global health and quality of life scale uses a 7-point scale scoring with anchors (1=very poor and 7=excellent); the other items are scored on a 4 point scale (1=not at all, 2=a little, 3= quite a bit, 4=very much).
Assessment of quality of life via the EORTC QLQ-BR42 questionnaire. | 3 years.
  Patient reported outcomes via the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Breast Cancer 42 (EORTC QLQ-BR42). It consists of 42 items that formed ten scales (Breast Symptoms, Body Image, Sexual Functioning, Arm Symptoms, Systemic Chemotherapy Side Effects, Hand/Feet Symptoms/Neuropathy, Skeletal Symptoms Scale, Endocrine Symptoms, Breast Satisfaction, Vaginal Symptoms) and 3 single items (Weight Gain, Sexual Enjoyment, and Future Perspective). The items are scored on a 4 point scale (1=not at all, 2=a little, 3= quite a bit, 4=very much).
Assessment of quality of life via the EQ-5D-5L questionnaire. | 3 years.
  Patient reported outcomes via the 5-level EuroQol-5D (EQ-5D-5L questionnaire). It consists of 5 health state dimensions: mobility, self-care, usual activities, pain, and anxiety. Each dimension is rated on a five-point scale from 1 (extreme problem) to 5 (no problem). It also includes a vertical visual analog scale with a graded scoring system: 0 represents the worst imaginable health status, while 100 represents the best.
Assessment of quality of life via the HADS questionnaire. | 3 years.
  Patient reported outcomes via the Hospital anxiety and depression scale (HADS). It is a 14 items questionnaire: 7 items related to anxiety and 7 items related to depression scored on a scale. Each item is rated on a 4-point Likert scale (0 = "not at all", 1 = "a little", 2 = "quite a bit", and 3 = "very much"), with higher scores indicating more distress.
Assessment of quality of life via the FCRI questionnaire. | 3 years.
  Patient reported outcomes via the Fear of Cancer Recurrence Inventory (FCRI). The scale is assessed using a 5-point Likert scale, where level 0 indicates "never or not at all" and level 4 indicates "a lot or always".
AE | 3 years.
  Incidence and severity of adverse events
Cost-Utility Analysis | 3 years.
  Measured by incremental cost-effectiveness ratio (ICER), expressed as the cost per quality-adjusted life year (QALY) gained.

OTHER OUTCOMES:
Biomarker | 3 years (before and after therapy).
  Compare the differences in immune cell proportion, PD-1 saturation and other aspects among blood and tissue samples in both arms to identify biomarkers that may predict treatment outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Breast Tumor Center, Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong, China